CLINICAL TRIAL: NCT01495819
Title: Nicotine Reinforcement and Aversion in Young Adult Light Smokers
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Mehmet Sofuoglu, Principle Investigator, Yale University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1010007514; 1R01DA042528-01 (NIH)
Record Dates: First submitted 2011-12-07; First posted 2011-12-20 (Estimated); Results first posted 2021-08-31 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Nicotine Addiction
Keywords: Nicotine; smokers; vitals associated with smoking
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Sodium Chloride; Nicotine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nicotine (Active Comparator): subjects will be randomly assigned to one of the five doses of nicotine (0.0125, 0.025, 0.0.5, 0.1 and 0.2 mg/70 kg or about 0.18, 0.36, 0.7, 1.4 and 2.8 µg/kg). At the beginning of each experimental session, subjects will first sample the assigned nicotine dose and placebo (saline) condition that are randomly labeled as A or B. which may be nicotine or saline. This procedure will allow subjects to sample the nicotine and saline that will be available during that session. In addition, subjective and physiological responses to the sample nicotine dose and saline will be assessed.
  Interventions: Drug: Nicotine
- Saline (Placebo Comparator): Subjects will have sample A and B, one being nicotine and one being saline. The doses will be blinded from PI, subject and staff. The subject must choose A or B for the next ten choices.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Saline — 5cc's of saline give at least once.
  Other Names: Placebo
  Arms: Saline
Drug: Nicotine — (0.0125, 0.025, 0.0.5, 0.1 and 0.2 mg/70 kg or about 0.18, 0.36, 0.7, 1.4 and 2.8 µg/kg).
  Other Names: IV nicotine
  Arms: Nicotine

SUMMARY:
The proposed study will examine the threshold for nicotine self-administration (NSA) using five different nicotine doses in young adult male and female non-dependent smokers (light and intermittent smokers or LITS). We propose a double-blind, placebo-controlled study that will enroll 195 individuals, targeting a total of 72 completers (36 male and 36 females). In each of the five experimental sessions, smokers will be randomly assigned to one of the five doses of nicotine (0.0125, 0.025, 0.05, 0.1 and 0.2 mg/70 kg). The highest dose, 0.2 mg/70 kg, corresponds to nicotine delivered by about one or two puffs of a cigarette. At the beginning of each experimental session, smokers will sample the assigned both the nicotine dose for that experimental session, and the placebo (saline) dose, followed by the opportunity to choose between nicotine and placebo for a total of ten choices over a 150-minute period. The main outcomes will be threshold dose (the minimum dose of nicotine that is self-administered more than placebo) and the slope of dose-response for nicotine self-administration (changes in nicotine self-administration per unit change in nicotine dose). We will also collect measures of nicotine intake (cotinine), nicotine clearance (3-hydroxycotinine (3-HC) / cotinine), and self-report drug effects

DETAILED DESCRIPTION:
Aim #1: To assess the threshold reinforcing dose and dose-effect curve for IV NSA at low doses in young adult LITS.

Hypothesis #1A: The threshold reinforcing doses for IV NSA will be between 0.0125 to 0.1 mg/70 kg.

Hypothesis #1B: The dose-effect curve for NSA will differ between males and females with relatively flat curve in female smokers.

Aim #2: To assess the threshold and dose-effect curve for the positive and negative/aversive subjective effects of IV nicotine at low doses and its relationship to nicotine reinforcement.

Hypothesis #2 A: The threshold for the positive effects will be between 0.0125 to 0.1 mg/70 kg, for the negative/aversive effect it will be ≥ 0.1 mg/70 kg.

Hypothesis #2B: Nicotine reinforcement will be positively correlated with the positive and negatively correlated with the negative/aversive subjective effects of IV nicotine.

Exploratory Aims: To examine the influence of nicotine clearance rate on nicotine reinforcement threshold and dose-effect curve.

ELIGIBILITY:
Inclusion criteria: 1) Female and male smokers, aged 18 to30 years, who have been smoking for at least a year, and a life-time consumption of at least 100 cigarettes; 2) smoke more frequently than once a week and ≤5 cpd; 3) FTND score <3 indicating no or minimal evidence for nicotine dependence; 4) urine cotinine levels >100 ng/mL indicating smoking status and a level <1000 mg/mL consistent with nicotine intake of LITS; 5) not seeking treatment at the time of the study for nicotine dependence; 6) in good health as verified by medical history, screening examination, and screening laboratory tests; 7) for women, not pregnant as determined by pregnancy screening, nor breast feeding, and using acceptable birth control methods.

Exclusion criteria: 1) history of major medical illnesses that the physician investigator deems as contraindicated for the subject to be in the study; 2) requirement of any form of regular psychotropic medication (antidepressants, antipsychotics, or anxiolytics) or psychiatric diagnosis and treatment for psychiatric disorders including major depression, bipolar disorder, schizophrenia in the past 6 months; and 3) current dependence to alcohol or any other recreational or prescription drugs and; 4) daily use of smokeless tobacco products or exclusive daily use of e-cigarettes (non-daily users will be included).

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2017-01-04 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Sofuoglu, M.D,Ph.D., Principal Investigator — Yale University
Locations (1):
- Department of Veterans Affairs, West Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] MacLean RR, Eid T, Parida S, Gueorguieva R, DeVito EE, Sofuoglu M. Threshold for the pleasurable effects of nicotine are lower than its reinforcing effects during self-administration. Exp Clin Psychopharmacol. 2023 Feb;31(1):37-45. doi: 10.1037/pha0000556. Epub 2022 Mar 7. PMID 35254839

RESULTS

PARTICIPANT FLOW:
Groups:
- Study Participants: subjects will be randomly assigned to one of the five doses of nicotine (0.0125, 0.025, 0.0.5, 0.1 and 0.2 mg/70 kg or about 0.18, 0.36, 0.7, 1.4 and 2.8 µg/kg). At the beginning of each experimental session, subjects will first sample the assigned nicotine dose and placebo (saline) condition that are randomly labeled as A or B. which may be nicotine or saline. This procedure will allow subjects to sample the nicotine and saline that will be available during that session. In addition, subjective and physiological responses to the sample nicotine dose and saline will be assessed.
Period: Overall Study
Arm/Group | Study Participants
Started | 34
Nicotine 0.0125 | 31
Nicotine 0.025 | 32
Nicotine 0.05 | 33
Nicotine 0.1 | 31
NIcotine 0.2 | 33
Completed | 30
Not Completed | 4

BASELINE CHARACTERISTICS:
Groups:
- Study Participants: In this crossover study, all participants received all 5 treatments, including placebo.
Arm/Group | Study Participants
Number analyzed (Participants) | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.7 (3.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 30
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 26
  White | 4
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 34
FTND [Mean (Standard Deviation); unit: units on a scale] — Participants in the study had to have a Fagerstrom Test of Nicotine Dependence (FTND) score < 3 indicating no or minimal evidence for nicotine dependence.
  Score range is 0-10 Score Interpretation 0-2 Very low level of dependence on nicotine. 3-4 Low level of dependence on nicotine. 5 Medium level of dependence on nicotine. 6-7 High level of dependence on nicotine. 8-10 Very high level of dependence on nicotine.
  units on a scale | 1.6 (1.3)
Average cigarettes per day [Mean (Standard Deviation); unit: cigarettes per day] | 4.5 (1.1)
Years of smoking [Mean (Standard Deviation); unit: years] | 8.7 (4.4)
Serum cotinine level [Mean (Standard Deviation); unit: ng/mL] — Cotinine extracted from blood serum samples.
  ng/mL | 137.4 (104.0)

OUTCOME MEASURES:

1. Primary Outcome: DEQ - Pleasurable
Description: The Drug Effects Questionnaire (DEQ) ratings subscale that measures the pleasurable effects was used. I The minimum score is zero with the maximum score of a 100millimeters.
  The higher the score means the more pleasurable.
Time Frame: Up to 10 Minutes
Population: Thirty four subject were randomized, 4 didn't complete all five test sessions, the sessions that were completed were analyzed.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Study Participants
Number analyzed (Participants) | 34
score on a scale
  Placebo | 2.14 (0.20)
  0.0125: number analyzed (Participants) | 31
  0.0125 | 2.05 (0.26)
  0.025: number analyzed (Participants) | 32
  0.025 | 1.98 (0.26)
  0.05: number analyzed (Participants) | 33
  0.05 | 2.37 (0.25)
  0.1: number analyzed (Participants) | 31
  0.1 | 2.67 (0.26)
  0.2: number analyzed (Participants) | 33
  0.2 | 3.24 (0.26)

2. Primary Outcome: DEQ - Aversive
Description: The DEQ is measured using millimeters. The minimum score is zero with the maximum score of a 100millimeters. rug Effects Questionnaire (DEQ) ratings subscale that measures the aversive effects was used. The higher the score means more aversive.
Time Frame: Up to 10 Minutes
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Study Participants
Number analyzed (Participants) | 34
score on a scale
  Placebo | 1.30 (0.20)
  0.0125: number analyzed (Participants) | 31
  0.0125 | 1.26 (0.22)
  0.025: number analyzed (Participants) | 32
  0.025 | 1.50 (0.22)
  0.05: number analyzed (Participants) | 33
  0.05 | 1.21 (0.22)
  0.1: number analyzed (Participants) | 31
  0.1 | 1.22 (0.22)
  0.2: number analyzed (Participants) | 33
  0.2 | 1.37 (0.22)

3. Primary Outcome: DEQ - Stimulatory
Description: The Drug Effects Questionnaire (DEQ) ratings subscale that measures the stimulatory effects was used.
  DEQ is measured using millimeters. The minimum score is zero with the maximum score of a 100millimeters. The higher the score means more stimulation.
Time Frame: Up to10 Minutes
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Study Participants
Number analyzed (Participants) | 34
score on a scale
  Placebo | 1.95 (0.20)
  0.0125: number analyzed (Participants) | 31
  0.0125 | 1.82 (0.25)
  0.025: number analyzed (Participants) | 32
  0.025 | 1.85 (0.25)
  0.05: number analyzed (Participants) | 33
  0.05 | 2.29 (0.24)
  0.1: number analyzed (Participants) | 31
  0.1 | 2.76 (0.25)
  0.2: number analyzed (Participants) | 33
  0.2 | 3.18 (0.24)

ADVERSE EVENTS:
Time Frame: Each subject participated in five laboratory sessions. Each participant were evaluated for adverse events each day for the five laboratory sessions
Groups:
- Saline: In this crossover study, all participants received all 5 treatments, including placebo.
- Nicotine 0.0125: All participants received 0.0125
- Nicotine 0.025: All participants received 0.025
- Nicotine 0.05: All participants received 0.05
- Nicotine 0.1: All Participants received 0.1
- Nicotine 0.2: All participants received 0.2
Arm/Group | Saline | Nicotine 0.0125 | Nicotine 0.025 | Nicotine 0.05 | Nicotine 0.1 | Nicotine 0.2
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/31 | 0/32 | 0/33 | 0/31 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/31 | 0/32 | 0/33 | 0/31 | 0/33
Other Adverse Events (participants affected / at risk) | 0/34 | 0/31 | 0/32 | 0/33 | 0/31 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-14): https://cdn.clinicaltrials.gov/large-docs/19/NCT01495819/Prot_SAP_000.pdf